CLINICAL TRIAL: NCT07321535
Title: Huangjing Yangji Formula Combined With Resistance Training for Sarcopenia: a Multicenter, Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Huangjing Yangji Formula Combined With Resistance Training for Sarcopenia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wangjing Hospital, China Academy of Chinese Medical Sciences (Other)
Collaborators: The First Affiliated Hospital of Tianjin University of Traditional Chinese Medicine (Other); Hunan University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WJEC-KT-2025-040-P001
Record Dates: First submitted 2025-12-21; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Sarcopenia
Keywords: traditional Chinese medicine; resistance training; randomized controlled trial; multicenter trial
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Huangjing Yangji Formula + Training (Experimental): Participants in this group will take "Huangjing Yangji Formula" granules orally. The formula consists of Polygonati rhizoma (Huangjing) 15g, Codonopsis radix (Dangshen) 10g, Rehmanniae radix praeparata (Shudi) 9g, Angelica sinensis radix (Danggui) 6g, Cistanches herba (Roucongrong) 9g, Lycii fructus (Gouqi) 12g, Poria (Fuling) 9g, and Crataegi fructus (Shanzha) 6g per daily dose. The granules are taken twice daily, 30 minutes after meals, for a total treatment period of 3 months. Additionally, all participants in this group will simultaneously complete the standardized elastic band resistance training program 3 times per week for 3 months.
  Interventions: Drug: Huangjing Yangji Formula Granules; Behavioral: Standardized Elastic Band Resistance Training Program
- Placebo + Training (Placebo Comparator): Participants in this group will take matched placebo granules orally. The placebo is designed to be identical to the investigational "Huangjing Yangji Formula" granules in appearance, color, odor, packaging, and solubility, but it contains no active herbal components. The placebo granules are taken twice daily, 30 minutes after meals, for a total treatment period of 3 months. Additionally, all participants in this group will simultaneously complete the identical standardized elastic band resistance training program 3 times per week for 3 months.
  Interventions: Drug: Placebo Granules for Huangjing Yangji Formula; Behavioral: Standardized Elastic Band Resistance Training Program

INTERVENTIONS:
Drug: Huangjing Yangji Formula Granules — Investigational herbal granule formulation. Each daily dose contains: Polygonati rhizoma (Huangjing) 15g, Codonopsis radix (Dangshen) 10g, Rehmanniae radix praeparata (Shudi) 9g, Angelica sinensis radix (Danggui) 6g, Cistanches herba (Roucongrong) 9g, Lycii fructus (Gouqi) 12g, Poria (Fuling) 9g, and Crataegi fructus (Shanzha) 6g. Administered orally as granules dissolved in water, twice daily (30 minutes after meals), for a period of 3 months.
  Arms: Huangjing Yangji Formula + Training
Drug: Placebo Granules for Huangjing Yangji Formula — Matched placebo granules. This preparation is specifically designed to be indistinguishable from the active "Huangjing Yangji Formula Granules" in terms of appearance, color, odor, packaging, and solubility. It contains no pharmacologically active herbal components. Administered orally in the same manner (twice daily, 30 minutes after meals) for 3 months.
  Arms: Placebo + Training
Behavioral: Standardized Elastic Band Resistance Training Program — A structured, progressive resistance training program using elastic bands. Participants train 3 times per week for 3 months. Each 60-minute session includes warm-up, 10 core strength exercises (e.g., standing row, leg extension, bridge), and cool-down. Intensity is progressively increased from low (approximately 40-60% of 1-RM) to medium-high (approximately 60-80% of 1-RM) resistance. Sessions are supervised once weekly, with twice-weekly home-based sessions.

SUMMARY:
The goal of this clinical trial is to learn if a traditional Chinese medicine formula called "Huangjing Yangji Formula," combined with elastic band resistance training, works better than exercise alone to improve physical function and muscle strength in older adults with sarcopenia (age-related muscle loss). The main questions it aims to answer are:

Does the combined treatment improve participants' overall physical performance scores more than exercise with a placebo?

Does it lead to better outcomes in walking speed, balance, muscle strength, body composition, nutrition, mood, sleep, and overall quality of life?

Researchers will compare two groups. One group will take the real Huangjing Yangji Formula granules and do the standardized elastic band resistance training. The other group will take placebo granules (a look-alike mixture with no active medicine) and do the same training.

Participants will:

Take the assigned granules twice daily for 3 months.

Complete a standardized elastic band exercise program 3 times per week for 3 months (with both group and home sessions).

Attend three assessment visits (at the start, after 3 months, and 1 month after treatment) for tests and questionnaires.

Provide blood samples at the start and after 3 months for routine safety tests and special muscle health markers.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled clinical trial evaluating the efficacy and safety of the traditional Chinese medicine prescription"Huangjing Yangji Formula" combined with elastic band resistance training for treating sarcopenia adults. A total of 106 eligible participants will be recruited from three tertiary hospitals in China and randomly assigned (1:1) to two groups. The experimental group will receive Huangjing Yangji Formula granules (composition: Polygonati rhizoma 15g, Codonopsis radix 10g, Rehmanniae radix praeparata 9g, Angelica sinensis radix 6g, Cistanches herba 9g, Lycii fructus 12g, Poria 9g, Crataegi fructus 6g) orally twice daily for 3 months. The control group will receive matched placebo granules on the same schedule. Both groups will simultaneously perform a standardized elastic band resistance training program 3 times per week for 3 months. The primary outcome is the change in the Short Physical Performance Battery (SPPB) score from baseline to 3 months. Secondary outcomes include physical function (gait speed, Timed Up and Go test, handgrip strength, Tinetti POMA score), body composition, frailty (FRAIL scale), activities of daily living (Barthel Index), nutrition (MNA-SF), psychological status (GDS-30, PSQI), quality of life (SF-12), TCM syndrome score, and serum biomarkers of inflammation and muscle metabolism. Outcome assessments occur at baseline, 3 months, and at a 1-month follow-up (4 months), except for serum biomarkers measured only at baseline and 3 months. Safety will be monitored through laboratory tests and adverse event recording.

ELIGIBILITY:
Inclusion Criteria:

* Meets the diagnostic criteria for sarcopenia according to the Asian Working Group for Sarcopenia (AWGS) 2025 consensus, defined as the co-presence of:

Low Muscle Mass: Appendicular skeletal muscle index (ASMI) measured by multi-frequency bioelectrical impedance analysis (BIA) below the following thresholds:

Ages 50-64: <7.6 kg/m² for men, <5.7 kg/m² for women. Ages ≥65: <7.0 kg/m² for men, <5.7 kg/m² for women.

Low Muscle Strength: Handgrip strength below the following thresholds:

Ages 50-64: <34 kg for men, <20 kg for women. Ages ≥65: <28 kg for men, <18 kg for women.

* Meets the Traditional Chinese Medicine (TCM) pattern diagnosis criteria for Spleen-Kidney Deficiency Syndrome, characterized by:

Primary Symptoms: Muscle wasting, general fatigue, soreness and weakness of the lower back and knees.

Secondary Symptoms: Poor appetite, abdominal distension, loose or chronic diarrhea, dizziness, poor memory. Tongue presentation: pale and swollen tongue with tooth marks, white and glossy coating. Pulse: deep, thin, and weak.

* Aged between 50 and 75 years.
* Willing and able to provide written informed consent personally or via a legal guardian.

Exclusion Criteria:

* Secondary sarcopenia due to specific diseases (e.g., active malignancy, hyperthyroidism, severe hepatic or renal dysfunction).
* Presence of severe or uncontrolled cardiovascular disease, consumptive diseases (e.g., cancer), active infections, or severe osteoporosis.
* Diagnosis of Alzheimer's disease, psychiatric disorders, or other cognitive/mental impairments that would hinder cooperation with the trial procedures.
* Inability to perform activities of daily living or walk independently; or presence of motor dysfunction due to joint deformities, prolonged bed rest, fractures, or other reasons that would preclude safe participation in resistance training.
* Known contraindications to the ingredients of the investigational herbal formula or allergy to the materials of the elastic bands.
* Use of medications known to affect muscle metabolism (e.g., corticosteroids, muscle relaxants) within the past 3 months.
* Participation in any other interventional clinical trial within the past 3 months.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Short Physical Performance Battery (SPPB) Score | Baseline, 3 months, and 4 months (1-month follow-up).
  The SPPB is a composite score ranging from 0 to 12 that assesses lower extremity physical function. It combines three tests: standing balance, 4-meter walking speed, and time to complete five chair stands. Scores are interpreted as: 0-3 (severe limitation), 4-6 (mild limitation), 7-9 (normal function), and 10-12 (excellent function). A higher score indicates better physical performance.

SECONDARY OUTCOMES:
4-Meter Walking Speed | Baseline, 3 months, and 4 months (1-month follow-up).
  Usual walking speed (in meters per second) assessed over a 4-meter course. Participants are instructed to walk at their normal, comfortable pace. The average speed of two trials is calculated and used for analysis. This is a key measure of mobility and functional capacity.
Timed Up and Go Test (TUG) | Baseline, 3 months, and 4 months (1-month follow-up).
  Time (in seconds) required to stand up from a standard armchair, walk 3 meters at a usual pace, turn around, walk back, and sit down again. The test is performed twice, and the shorter time of the two trials is recorded. It is a widely used measure of functional mobility and fall risk.
Handgrip Strength | Baseline, 3 months, and 4 months (1-month follow-up).
  Maximal isometric strength of the dominant hand, measured in kilograms (kg) using a handheld dynamometer (handgrip). The participant is seated with the forearm supported. Three trials are performed, and the highest value is recorded as the outcome. It is a standard measure of overall muscle strength.
Tinetti Performance-Oriented Mobility Assessment (POMA) | Baseline, 3 months, and 4 months (1-month follow-up).
  Total score on the POMA, a standardized tool to assess balance and walking ability. It consists of a Balance subscale (9 items, score 0-16) and a Gait subscale (7 items, score 0-12). The total score ranges from 0 to 28, with a higher score indicating better mobility and lower fall risk. Scores are interpreted as: ≤18 (high fall risk), 19-24 (moderate fall risk), ≥25 (low fall risk).
Appendicular Skeletal Muscle Index (ASMI) | Baseline, 3 months, and 4 months (1-month follow-up).
  The appendicular skeletal muscle mass (sum of muscle mass in both arms and legs) measured in kilograms (kg) using a multi-frequency BIA device (InBody 770C), divided by the square of height in meters to yield ASMI in kg/m².
Lean Body Mass | Baseline, 3 months, and 4 months (1-month follow-up).
  Lean body mass measured in kilograms (kg) using a multi-frequency bioelectrical impedance analysis (BIA) device (InBody 770C).
Fat Mass | Baseline, 3 months, and 4 months (1-month follow-up).
  Fat mass measured in kilograms (kg) using a multi-frequency bioelectrical impedance analysis (BIA) device (InBody 770C).
Body Fat Percentage | Baseline, 3 months, and 4 months (1-month follow-up).
  Body fat percentage measured in percent (%) using a multi-frequency bioelectrical impedance analysis (BIA) device (InBody 770C).
Body Mass Index (BMI) | Baseline, 3 months, and 4 months (1-month follow-up).
  Body Mass Index calculated as weight in kilograms divided by height in meters squared (kg/m²). Weight and height are obtained using a multi-frequency bioelectrical impedance analysis (BIA) device (InBody 770C).
FRAIL Scale Score | Baseline, 3 months, and 4 months (1-month follow-up).
  Total score on the FRAIL scale, a brief screening tool based on the frailty phenotype. It assesses five components: Fatigue, Resistance (difficulty climbing stairs), Ambulation (difficulty walking), Illnesses (number of comorbidities), and Loss of weight. Each component present scores 1 point. Total scores range from 0 to 5 and are interpreted as: 0 (robust/no frailty), 1-2 (pre-frail), and ≥3 (frail).
Barthel Index Score | Baseline, 3 months, and 4 months (1-month follow-up).
  Total score on the Barthel Index, a measure of independence in performing basic activities of daily living (ADL). It assesses 10 items: feeding, bathing, grooming, dressing, bowel control, bladder control, toilet use, bed-chair transfer, ambulation, and stair climbing. Each item is scored 0, 5, 10, or 15 based on the level of assistance required. Total scores range from 0 to 100 and are interpreted as: 0-20 (total dependence), 25-45 (severe dependence), 50-70 (moderate dependence), 75-95 (mild dependence), 100 (complete independence).
Geriatric Depression Scale (GDS) Score | Baseline, 3 months, and 4 months (1-month follow-up).
  Total score on the 30-item GDS, a self-report measure designed specifically to assess depressive symptoms, focusing on mood and cognition while minimizing somatic items. Scores range from 0 to 30. A total score of ≥11 indicates the presence of depressive symptoms, with scores of 11-20 suggesting mild depression and scores of 21-30 suggesting moderate to severe depression.
Mini Nutritional Assessment - Short Form (MNA-SF) Score | Baseline, 3 months, and 4 months (1-month follow-up).
  Total score on the MNA-SF, a 6-item screening tool used to assess nutritional status or risk of malnutrition. Total scores range from 0 to 14 and are interpreted as: 12-14 (normal nutritional status), 8-11 (at risk of malnutrition), and 0-7 (malnourished).
Pittsburgh Sleep Quality Index (PSQI) Score | Baseline, 3 months, and 4 months (1-month follow-up).
  Global score on the PSQI, a 19-item self-rated questionnaire assessing sleep quality and disturbances over the past month. The score encompasses seven components. Total scores range from 0 to 21, interpreted as: 0-5 (good sleep quality), 6-10 (mild sleep disturbance), 11-15 (moderate sleep disturbance), and 16-21 (severe sleep disturbance).
12-Item Short Form Health Survey (SF-12) score | Baseline, 3 months, and 4 months (1-month follow-up).
  Scores on the SF-12, a shortened version of the SF-36 used to efficiently assess health-related quality of life. It yields two summary scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). Both are standardized scores, with higher values indicating better physical or mental health-related quality of life.
Serum Biomarker Levels | Baseline and 3 months of intervention.
  Fasting venous blood samples will be collected, processed within 30 minutes, and stored for batch analysis. Levels of the following biomarkers will be quantified using standard methods: inflammatory markers (Tumor Necrosis Factor-alpha, Interleukin-6, Interleukin-1beta), muscle metabolism markers (Irisin, Myostatin), and metabolic hormones (25-Hydroxyvitamin D, Insulin-like Growth Factor-1, Growth Hormone).
Traditional Chinese Medicine (TCM) Syndrome Score | Baseline, 3 months, and 4 months (1-month follow-up).
  The TCM syndrome score is assessed according to the《Guiding Principles for Clinical Research of New Chinese Medicines》. It evaluates three primary symptoms (muscle wasting, general fatigue, soreness and weakness of the lower back) and five secondary symptoms (poor appetite, abdominal distension, loose stools, dizziness, forgetfulness). Primary symptoms are scored 0 (none), 2 (mild), 4 (moderate), or 6 (severe); secondary symptoms are scored 0 (none), 1 (mild), 2 (moderate), or 3 (severe). The total score is the sum of all items, with a higher score indicating more severe symptoms. Efficacy is categorized based on the percentage reduction in the total score after treatment: ≥70% (markedly effective), 30-69% (effective), <30% (ineffective).

CONTACTS AND LOCATIONS:
Overall Officials: Xu Wei, Ph.D., Principal Investigator — Wangjing Hospital, China Academy of Chinese Medical Sciences
Locations (3):
- China (3):
  - Wangjing Hospital, China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Hunan University of Chinese Medicine, Changsha, Hunan
  - The First Affiliated Hospital of Tianjin University of Traditional Chinese Medicine, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared publicly due to the need to protect participant privacy and in accordance with the data management policies of the participating hospitals in this multicenter trial.